CLINICAL TRIAL: NCT02155855
Title: Effectiveness of and Satisfaction With Remote Blood Glucose Monitoring and Telemedicine for Adolescents With Insulin-dependent Diabetes
Brief Title: Telemedicine for Adolescents With Insulin-dependent Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: L14-037
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes, home glucose monitor, upload, cloud
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): Telemedicine group will test blood glucose at least 4 times a day Each time the meter time-stamps the reading. All meter readings will upload to the cloud via "Myglucohealth" website, where they can be accessed by caregivers, including providers and parents. Parents will be notified by device about the blood glucose testing results. Provider will set device to alert patient or patient's family or send alerts if uploaded numbers are outside an identified range (<70 mg/dL > 300 mg/dL). As per the standard of care, parents are trained to administer sugar containing liquids, or inject extra insulin for hyperglycemia correction. Parents will be encouraged to contact study personnel if they are concerned about the diabetes control. Study personnel will access home blood glucose monitor data, and provide insulin dosing advice. Parents will be asked to upload blood glucose readings prior to each visit.
  Interventions: Other: Telemedicine
- Control (Active Comparator): Control Subjects will continue routine care which requires blood glucose testing at least 4 times a day. Parents will use customary ways to communicate (pager, email, fax or phone) with the Diabetes team, if they are concerned about glycemic control..
  Interventions: Other: Control

INTERVENTIONS:
Other: Telemedicine — Study group will test blood glucose at least 4 times a day Each time the meter timestamps the reading. All meter readings will upload to the cloud via Myglucohealth website, where they can be accessed by caregivers, including providers and parents. Parents will be notified by device about the blood glucose testing results. Provider will set device to alert patient or patient's family or send alerts if uploaded numbers are outside an identified range (<70 mg/dL > 300 mg/dL). As per the standard of care, parents are trained to administer sugar containing liquids, or inject extra insulin for hyperglycemia correction. Parents will be encouraged to contact study personnel if they are concerned about the diabetes control. Study personnel will access home blood glucose monitor data, and provide insulin dosing advice. Parents will be asked to upload blood glucose readings prior to each visit.
  Arms: Telemedicine
Other: Control — Routine care
  Arms: Control

SUMMARY:
Investigators hope that providing patients and families with additional ways of communication with the diabetes care team will improve diabetes control.

DETAILED DESCRIPTION:
Study Group Study group will be asked to test blood glucose at least 4 times a day Each time the study subject takes a meter reading the meter time-stamps the reading. All meter readings will upload to the cloud via" Myglucohealth" website, where they can be accessed by caregivers, including providers and parents. Device will be programmed to coax patients when readings are due. Parents will be notified by device about the blood glucose testing results. Provider will set device to alert patient or patient's family if patient has not yet tested or uploaded a test or send alerts to parent if uploaded numbers are outside an identified range (<70 mg/dL > 300 mg/dL). As per the standard of care, parents are trained to administer sugar containing liquids, or inject extra insulin for hyperglycemia correction. Parents will be encouraged to contact study personnel if they are concerned about the diabetes control. Study personnel will access home blood glucose monitor data, and provide insulin dosing advice. Parents will be asked to upload blood glucose readings prior to each visit.

Control group Subjects will continue routine care which requires blood glucose testing at least 4 times a day. Parents will use customary ways to communicate (pager, email, fax or phone) with the Diabetes team, if they are concerned about glycemic control..

Study group will have two virtual visits (months 3 and 6) Control group will have all quarterly visits in person. A laptop will be used for virtual visits and will be set up with the help of the TTUHSC Information Technology Security Officer.

ELIGIBILITY:
Inclusion Criteria:

-- Age 10-18 years

* Multiple daily injections regimen
* Duration of diabetes > 12 months
* HbA1c > 7%
* Lives outside of Lubbock
* Committed to visit schedule

Exclusion Criteria:

* Foster care or residential facility
* Psychiatric illness
* Developmental delay
* Reading at < 4th grade level
* Pregnancy
* Known seizure disorder

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c | 12 months
  As an indicator of diabetes control

SECONDARY OUTCOMES:
Frequency of contact with diabetes care team | 12 months
  To see if tele-communication is used more than the conventional (phone, FAX)

CONTACTS AND LOCATIONS:
Overall Officials: Daina Dreimane, MD, Principal Investigator — TTUHSC School of Medicine
Locations (1):
- TTUHSC Pediatric Clinic, Lubbock, Texas, United States